CLINICAL TRIAL: NCT04721769
Title: Endoscopic Strip Craniectomy for Treatment of Isolated, Non-syndromic Sagittal Craniosynostosis
Brief Title: Endoscopic Strip Craniectomy for Treatment of Sagittal Craniosynostosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, David Bauer, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-48130
Record Dates: First submitted 2021-01-06; First posted 2021-01-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Craniosynostosis, Sagittal
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Intervention Model Description: We have two patient groups. Group 1: Endoscopic strip craniectomy with the use of lateral osteotomies. Group 2: Endoscopic strip craniectomy without the use of lateral osteotomies.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and guardians of participants will not know which arm the participant is randomized to. Regarding care providers, only care providers performing the surgery will be privy to information regarding which arm the patient is randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopic strip craniectomy with the use of lateral osteotomies (Active Comparator): Patients will have lateral osteotomies incorporated into their surgical procedure following suturectomy of the fused sagittal suture.
  Interventions: Procedure: Endoscopic strip craniectomy (with lateral osteotomies) with post-operative helmet therapy
- Endoscopic strip craniectomy without the use of lateral osteotomies (Experimental): Patients will NOT have lateral osteotomies incorporated into their surgical procedure following suturectomy of the fused sagittal suture.
  Interventions: Procedure: Endoscopic strip craniectomy (without lateral osteotomies) with post-operative helmet therapy

INTERVENTIONS:
Procedure: Endoscopic strip craniectomy (with lateral osteotomies) with post-operative helmet therapy — Endoscopic strip craniectomy is a surgical procedure performed to remove pathologic bone of the calvarium that includes the fused suture. Lateral osteotomies, also known as barrel-stave osteotomies, are performed by some surgeons because of their perceived benefit in regard to cranial expansion. Following surgery, orthotic helmet therapy is performed in order to mold the calvarium with the goals of optimizing contour.
  Other Names: Endoscopic suturectomy (with barrel-stave osteotomies) with post-operative helmet therapy
  Arms: Endoscopic strip craniectomy with the use of lateral osteotomies
Procedure: Endoscopic strip craniectomy (without lateral osteotomies) with post-operative helmet therapy — Endoscopic strip craniectomy is a surgical procedure performed to remove pathologic bone of the calvarium that includes the fused suture. Lateral osteotomies, also known as barrel-stave osteotomies, are performed by some surgeons because of their perceived benefit in regard to cranial expansion. Following surgery, orthotic helmet therapy is performed in order to mold the calvarium with the goals of optimizing contour.
  Other Names: Endoscopic suturectomy (without barrel-stave osteotomies) with post-operative helmet therapy
  Arms: Endoscopic strip craniectomy without the use of lateral osteotomies

SUMMARY:
* Endoscopic strip craniectomy (ESC) with post-operative helmeting is the gold-standard treatment for isolated, non-syndromic sagittal craniosynostosis in children under 6 months of age as it is has been demonstrated to reduce perioperative morbidity when compared to more invasive procedures such as cranial vault remodeling. ESC is frequently performed with or without the use of lateral osteotomies with technical selection being largely based on surgeon preference.
* Previous studies have shown that there are no statistically significant differences in cranial expansion or complications between the two procedure variants; however, these studies are retrospective in nature and do not account for aesthetic outcomes.
* The purpose of this study is to compare the efficacy of ESC with or without the use of lateral osteotomies in regard to cranial expansion and aesthetic outcomes for children treated with isolated, non-syndromic sagittal craniosynostosis. In addition, we seek to investigate if there are any observable changes in perioperative morbidity between the two procedures.

DETAILED DESCRIPTION:
* This prospective, randomized parallel study seeks to compare the efficacy of ESC with or without the use of lateral osteotomies in regard to cranial expansion and aesthetic outcomes for children treated with isolated, non-syndromic sagittal craniosynostosis.
* Both arms of the study will undergo standard care throughout their participation which includes preoperative & postoperative measurements of cephalic index using the STARscanner© (Orthomerica products Inc.), preoperative & postoperative photographs, post-operative helmeting, and standard post-operative visits.
* Additional research-related activities include chart review. Primary outcomes include degree of cranial expansion at 1 year post-operatively.
* Secondary outcomes include aesthetic appearance at 1 year post-operatively (using a 5-point Likert scale) and a multitude of intraoperative clinical variables including estimated blood loss, instances of transfusion, instances of dural tear, instances of 30-day readmission, and instances of needing further surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients with isolated, non-syndromic sagittal craniosynostosis under 6 months of age who present to Texas Children's Hospital.

Exclusion Criteria:

* Patients who are unable to undergo endoscopic strip craniectomy by 6 months of age.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in cephalic index from preoperative measurement to postoperative measurement at 1 year of age | Pre-operatively (at recruitment) & post-operatively (at 1 year of age)
  The cephalic index is the ratio of maximal head width and length. Patients enrolled in the trial will undergo pre-operative and post-operative measurement of their cephalic index using the STARscanner© (Orthomerica products Inc.). Patients will undergo measurement at recruitment and at 1 year of age.

SECONDARY OUTCOMES:
Aesthetic outcome | post-operatively (at 1 year of age)
  The aesthetic appearance of the calvarium will be measured by participating surgeons using a 5-point Likert scale (1-5) with 1 being extremely satisfied with aesthetic outcome and 5 being extremely dissatisfied with aesthetic outcome. Surgeons that are aware of the participant's assignment are excluded from this portion of the study to minimize bias.
Operative length | during the intervention/procedure/surgery
  Length of operation from incision to closure
Estimated Blood loss | during the intervention/procedure/surgery
  Based on estimated volume of blood loss and perioperative changes in hemoglobin mass
Instance of transfusion | during the intervention/procedure/surgery
  Whether or not the participant received a blood transfusion intraoperatively or post-operatively
Amount of blood transfused | during the intervention/procedure/surgery
  Measured in mL/kg
Instance of dural tear | during the intervention/procedure/surgery
  Whether or not the patient experienced a dural tear during surgery
Instance of 30-day readmission | Day of procedure through 30 days post-operatively
  Whether or not a patient was readmitted to the hospital for complications related to their surgical procedure
Instance of needing further surgical correction | 1 year after surgery
  Whether or not the patient requires further surgical intervention to correct their calvarial defect.

CONTACTS AND LOCATIONS:
Overall Officials: David F Bauer, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wood BC, Ahn ES, Wang JY, Oh AK, Keating RF, Rogers GF, Magge SN. Less is more: does the addition of barrel staves improve results in endoscopic strip craniectomy for sagittal craniosynostosis? J Neurosurg Pediatr. 2017 Jul;20(1):86-90. doi: 10.3171/2017.1.PEDS16478. Epub 2017 Apr 14. PMID 28409698
- [Background] Nguyen DC, Farber SJ, Skolnick GB, Naidoo SD, Smyth MD, Kane AA, Patel KB, Woo AS. One hundred consecutive endoscopic repairs of sagittal craniosynostosis: an evolution in care. J Neurosurg Pediatr. 2017 Nov;20(5):410-418. doi: 10.3171/2017.5.PEDS16674. Epub 2017 Aug 25. PMID 28841109
- [Background] Fearon JA, Ditthakasem K, Herbert M, Kolar J. An Appraisal of the Cephalic Index in Sagittal Craniosynostosis, and the Unseen Third Dimension. Plast Reconstr Surg. 2017 Jul;140(1):138-145. doi: 10.1097/PRS.0000000000003422. PMID 28654600